CLINICAL TRIAL: NCT04040309
Title: Plasma Rich in Growth Factors Effectiveness for Myofascial Pain Treatment in Masticatory Muscles: a Randomized Controlled Clinical Trial
Brief Title: PRGF Effectiveness for Myofascial Pain Treatment in Masticatory Muscles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dovydas Šakalys, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE-10-10
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Myofascial Pain
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: The first group of patients will receive 1 ml PRGF 2nd fraction injections into the myofascial trigger point in the masseter muscle.
  The second group of patients will receive 1 ml 2% Lidocaine injections into the myofascial trigger point in the masseter muscle.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma rich in growth factors group (Experimental): Group of patients who will receive 1 ml of PRGF 2nd fractions injections into their trigger points in the masseter muscle.
  Interventions: Biological: PRGF injection
- Lidocaine group (Active Comparator): Group of patients who will receive 1 ml 2% Lidocaine injections into the myofascial trigger point in the masseter muscle.
  Interventions: Drug: Lidocaine injection

INTERVENTIONS:
Biological: PRGF injection — Plasma rich in growth factors will be prepared following the protocol described by E. Anitua. 9 ml of patients venous blood will be taken into one tube with 3,8% sodium citrate used as an anticoagulant. The blood then will be centrifuged (PRGF Centrifuge System, Biotechnology Institute, Vitoria, Spain) at room temperature for 8 min at 1800 rpm. After centrifugation 1 ml of 2nd plasma fraction will be collected by using a pipet. To activate plasma 10% calcium chloride will be used immediately before injecting plasma into the trigger point in the masseter muscle.
  Arms: Plasma rich in growth factors group
Drug: Lidocaine injection — 1 ml 2 % Lidocaine will be injected into the trigger point in the patient's masseter muscle.
  Arms: Lidocaine group

SUMMARY:
The investigators set up a randomized controlled clinical trial to evaluate the effectiveness of plasma rich in growth factors (PRGF) injections into the masseter muscle trigger points for myofascial pain treatment. The investigators also seek to compare PRGF injections effectiveness with local anesthetic injections.

Dry needling and local anesthetics injections release trigger point by disrupting the membranes of a tout band. However, the injected substance itself does not affect the pathophysiological mechanism of the trigger point.

It is known that the platelets release growth factors who can enhance muscle regeneration processes and moreover reduce chronic pain.

The investigators raised a hypothesis that PRGF injections into the trigger points in masseter muscle can be an effective treatment method for the myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Diagnosed myofascial pain syndrome in one side of the masseter muscle (diagnosis is based on diagnostic criteria described by Travell and Simons: 1) palpable taut band, 2) spot tenderness in a taut band, 3) pain recognition.
* Patients have never had injections into their masseter muscle.

Exclusion Criteria:

* Myofascial trigger points in other masticatory muscles.
* Head and neck region inflammations that causes pain.
* Temporomandibular joint pathology which causes pain.
* Trigeminal nerve neuralgia.
* Head and neck region oncological diseases.
* Myofascial trigger points in both sides of masseter muscles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Pain levels 2 weeks after the procedure: Visual analog scale | Patients pain levels will be measured 2 weeks after the procedure.
  Patients will evaluate pain by using the Visual analog scale from 0 to 10. Where 0 means no pain and 10 means the worst possible pain
Pain levels 4 weeks after the procedure: Visual analog scale | Patients pain levels will be measured 4 weeks after the procedure.
  Patients will evaluate pain by using the Visual analog scale from 0 to 10. Where 0 means no pain and 10 means the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Gintaras Januzis, PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- LUHS Kaunas clinics Department of Maxillofacial surgery, Kaunas, Lithuania